CLINICAL TRIAL: NCT01623284
Title: PiB PET Scanning in Speech and Language Based Dementias
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Keith A. Josephs, Consultant-Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-008772
Record Dates: First submitted 2012-06-07; First posted 2012-06-19 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: PPA; Primary Progressive Aphasia; Aphasia; Non-fluent Aphasia; Semantic Dementia; Apraxia of Speech; Primary Progressive Nonfluent Aphasia; Progressive Aphasia
Keywords: aphasia; apraxia of speech; language
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Aphasia, Broca; Frontotemporal Dementia; Apraxias; Primary Progressive Nonfluent Aphasia; Language | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PiB and FDG positron emission tomography (PET) (Experimental): All subjects will receive PiB and FDG PET diagnosis on approximately day 1 or day 2 of study to determine if they have beta-amyloid deposits in their brains.
  Interventions: Drug: C-11 PiB; Drug: F-18 FDG

INTERVENTIONS:
Drug: C-11 PiB — One time intravenous administration of 740 megabecquerel (MBq) of [N-methyl-11C]2-(4'-methylaminophenyl)-6-hydroxybenzothiazole (PiB) (range 370 - 740 MBq).
  Other Names: Pittsburgh Compound B
Drug: F-18 FDG — One time intravenous administration of 629 megabecquerel (MBq) of [18-F]-fluoro-deoxy-glucose (FDG) (range 555 - 740 MBq).
  Other Names: Fluorodeoxyglucose-18

SUMMARY:
The study is designed to determine whether there are clinical features that can be used as biomarkers to predict whether underlying Alzheimer's pathology is the cause of a speech and language based dementia. The primary hypothesis is that the proportion of patients who test positive for beta-amyloid deposition will vary across different speech and language based dementias.

DETAILED DESCRIPTION:
Speech and language based dementias (SLDs) (often referred to as primary progressive aphasias or PPA) are neurodegenerative diseases in which speech or language impairments are the most salient features of the disease and explain deficits in activities of daily living. Patients with SLDs may have poor grammar, prominent anomia, comprehension deficits, speech production and articulation problems, difficulty with repetition of words or sentences, word finding pauses, or a combination of all these features. The SLDs can be further divided into different subtypes. Up to 50% of patients with SLDs that go on to autopsy have shown Alzheimer type pathology where beta-amyloid deposition is observed; the rest have pathology consistent with frontotemporal lobar degeneration where beta-amyloid deposition is absent. Future disease modifying treatments that target beta-amyloid will most likely differ from treatments that do not target beta-amyloid. As a consequence, biomarkers are needed to differentiate patients with SLDs with and without beta-amyloid deposition.

Little research has been done to identify biomarkers that could differentiate patients with SLDs with and without beta-amyloid, mainly because the gold standard to identify the presence of beta-amyloid has been pathological examination, which does not always occur, and may not occur until more than 10 years after onset. The recent development of [N-methyl-11C]2-(4'-methylaminophenyl)-6-hydroxybenzothiazole also known as 11C Pittsburgh Compound B or PiB is a solution to this problem since PiB allows the in vivo detection of beta-amyloid. Unfortunately, PiB is very expensive.

The long term goal of our research is to develop a cost effective algorithmic approach to the evaluation and diagnosis of patients presenting with SLDs. The objective of the studies outlined in this proposal is to identify clinical, neuropsychological, or imaging biomarkers that are readily available, relatively inexpensive, and non-invasive that will allow the differentiation of patients with SLDs with and without beta-amyloid deposition. We will use PiB as an indicator of beta-amyloid pathology. Our proposal is predicated upon our strong preliminary data showing that clinical, neuropsychological and radiological features differ between patients with SLDs with and without beta-amyloid deposition. Our central hypothesis is that temporo-parietal lobe findings such as memory loss, visuospatial/perceptual impairment, parietal lobe atrophy on magnetic resonance imaging (MRI), and parietal lobe hypometabolism on [18-F]-fluoro-deoxy-glucose positron emission tomography (FDG-PET), will be associated with beta-amyloid deposition (PiB positive status). On-the-other hand, frontal lobe features, such as apraxia of speech and behavioral and executive dysfunction, as well as extrapyramidal features such as Parkinsonism, will be associated with absence of beta-amyloid deposition (PiB negative status). The rationale for examining these clinical-imaging relationships is that successful predictions will provide a solid scientific foundation for the ultimate development of a cost effective algorithm to guide the diagnosis of SLDs.

Patients found to be eligible and willing to enroll in this study will be asked to undergo a Neurologic Examination, a Speech Pathology Consultation, Neuropsychometric testing, an MRI scan, an FDG PET scan and a PiB PET scan of the brain. This will be done over a period of two days at the Mayo Clinic in Rochester, MN.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Has an informant/study partner who will be able to provide independent evaluation of functioning
* Speaks English as their primary language (including bilingual patients whose primary language is English)
* Fulfills diagnostic criteria for PPA (Primary Progressive Aphasia) or Progressive Apraxia of Speech
* Agrees to and is eligible to undergo MRI and PET scanning
* If woman of child bearing age, pt must agree to pregnancy test no more than 48 hours before the PET scans

Exclusion Criteria:

* Any concurrent illnesses that could account for speech and language deficits, such as:

  * traumatic brain injury, strokes and developmental syndromes
  * patients meeting criteria for another neurodegenerative disease (Alzheimer's Disease, Dementia with Lewy Bodies, behavioral variant frontotemporal dementia, progressive supranuclear palsy, corticobasal degeneration)
* Women who is pregnant or post-partum and breast-feeding
* Patients for which MRI is contraindicated (metal in head, cardiac pace maker, etc.), if there is severe claustrophobia, if there are conditions that may confound brain imaging studies (e.g. structural abnormalities, including subdural hematoma or intracranial neoplasm), or if they are medically unstable or are on medications that might affect brain structure or metabolism,(e.g. chemotherapy)
* Patient is mute (secondary to dysarthria only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2010-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with different speech and language based dementia (SLD) subtypes who have a [N-methyl-11C]2-(4'-methylaminophenyl)-6-hydroxybenzothiazole (PiB) positive positron emission tomography (PET) scan at presentation | Study entry, approximately day 1 or day 2 of study

SECONDARY OUTCOMES:
Percentage of patients who exhibit apraxia of speech as measured by the Apraxia of Speech Rating Scale at presentation | Study entry, approximately day 1 or day 2 of study
  Apraxia of Speech Rating Scale has been developed by the speech pathologists involved in this study, and has tested to be reliable. The scale ranges from 0-4; 0=apraxia of speech not present, 4=apraxia of speech nearly always evident and marked in severity.
Temporoparietal hypometabolism as shown on [18-F]-fluoro-deoxy-glucose positron emission tomography (FDG-PET) scan at presentation | Study entry, approximately day 1 or day 2 of study
Grey matter loss as shown on magnetic resonance imaging (MRI) at presentation | Study entry, approximately day 1 or day 2 of study

CONTACTS AND LOCATIONS:
Overall Officials: Keith A Josephs, M.D. MST, MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States